CLINICAL TRIAL: NCT05638412
Title: Investigating the Impact of JASPER Behavioral Therapy in Children With Down Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Carol Wilkinson, Assistant Professor, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P00043317
Record Dates: First submitted 2022-11-09; First posted 2022-12-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Down Syndrome
Keywords: Parent Coaching; Parent Education; Social Communication; Play Skills; Behavioral regulation; Development; Emotional regulation
MeSH Terms: conditions — Down Syndrome; Communication; Emotional Regulation | interventions — Activator Appliances

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JASPER Intervention Group (Experimental): Caregivers receiving the JASPER intervention will undergo weekly virtual 60-minute sessions for 10 weeks conducted via Zoom.
  The content of the intervention includes teaching and implementation of contingent responding and specific strategies to provide a high-quality response to children's communication, and play behaviors. Caregiver training is completed through review of pre-recorded videos of the caregiver-child dyad each week. The first half of each session will be dedicated to reviewing previous content and feedback on the play recording. The following half will consist of new material. The coaching support includes contingent responding, the parent is also taught to use specific strategies to provide a rich, high-quality response to children's communication, and play behaviors.
  Interventions: Behavioral: JASPER
- Psychoeducational Curriculum Group (Experimental): Caregivers receiving the 10 weekly psychoeducational curriculum modules will be provided with the resources via secure email and encouraged to engage with the material a self-directed manner.
  The psychoeducational modules will include written information about child development, communication and social interaction skills, behavioral principles for managing challenging behavior and strategies for teaching new skills. No direct caregiver-child mediated coaching will be provided. The content of the modules will include information about developmental milestones in this age group for children with DS, behavior management strategy recommendations, positive parenting materials, and materials on increasing engagement through play.
  Interventions: Behavioral: Psychoeducational Curriculum

INTERVENTIONS:
Behavioral: JASPER — JASPER is a therapist and caregiver-mediated intervention that (1) targets the foundations of social communication, (2) uses naturalistic behavioral strategies to increase the rate and complexity of social communication and (3) includes caregivers as implementers of the intervention to promote generalization across settings and to ensure maintenance. This intervention is individualized and centered around two key developmental domains critical for social communication function: joint engagement and joint attention.
  Arms: JASPER Intervention Group
Behavioral: Psychoeducational Curriculum — The psychoeducational modules will include written information about child development, communication and social interaction skills, behavioral principles for managing challenging behavior and strategies for teaching new skills. No direct caregiver-child mediated coaching will be provided. The material provided will be similar to what a pediatrician or developmental specialist may review as a part of routine care.
  Arms: Psychoeducational Curriculum Group

SUMMARY:
In this study, investigators will study the impact of a 1:1 caregiver coaching intervention using the JASPER (Joint Attention, Symbolic Play, Engagement, Regulation) behavioral therapy curriculum compared to a psychoeducational curriculum that will be provided to caregivers for self-directed learning. Investigators want to determine the impact of both interventions on the child's development and behavior, and caregiver implementation of strategies.

DETAILED DESCRIPTION:
Down syndrome (DS), the most common genetic cause of intellectual disability, can be associated with a wide range of developmental needs. Behavioral challenges are common, and can impact learning, overall achievement, relationships, inclusion in schools, and community integration.

The goal of this study is to determine whether JASPER (Joint Attention Symbolic Play Engagement and Regulation) can improve caregiver implementation of behavioral strategies, caregiver self-efficacy and confidence, and child development.

Participants will be randomized to receive either the JASPER intervention or a caregiver psychoeducational group. Participants in the JASPER intervention will receive 10 weekly virtual educational sessions utilizing JASPER therapy modules through 1:1 parent-child coaching sessions. Caregivers in the comparison group will receive 10 weekly modules containing a psychoeducational curriculum. The outcome measures will assess caregiver responsiveness, child joint engagement with caregiver, caregiver self-efficacy, and child behavior, language, and adaptive skills.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Trisomy 21
* Age 3-7 years
* Able to walk independently
* English speaking
* Caregiver able to complete either 1:1 virtual coaching sessions or psychoeducational behavioral curriculum

Exclusion Criteria:

* Mosaic Down syndrome
* Significant and uncorrected hearing and/or vision problems

Ages: 36 Months to 90 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Joint engagement and joint attention skills | 20 weeks
  Joint engagement and joint attention skills will be coded from Caregiver-Child Interaction (CCX) video recordings. The 15-minute CCX videos measure the amount of time that caregiver and child engage during a play session. The frequency of the child's engagement states will be coded using an Engagement State Coding Scheme to measure proportion of video during which child is maintaining Joint Engagement (shared engagement in a play routine).
Social communication skills | 20 weeks
  Social communication skills will be coded from Caregiver-Child Interaction (CCX) video recordings. The 15-minute CCX videos measure the amount of time that caregiver and child engage during a play session. A Social Communication Coding Scheme will measure the child's social communication skills. This coding scheme includes various social communication items and "Yes" or "No" codes to measure social communication skill development over time. Increasing answers of "Yes" indicate growth in social communication skills.
Caregiver use of behavioral strategies | 20 weeks
  The frequency with which caregivers use behavioral strategies will be collected from a weekly caregiver Behavioral Strategy Log.
Language, socialization, play, problem behavior, and adaptive skills | 20 weeks
  Language, socialization, play, problem behavior, and adaptive skills measured by a parent interview about development using the Vineland Adaptive Behavior Scales (VABS-III). Behavior frequency is measured on a range of 0=Never to 1=Sometimes to 2=Usually.
Socialization and play skills | 20 weeks
  Socialization and play skill development measured by the Play Assessment Questionnaire. The Play Assessment Questionnaire includes "Yes" or "No" items about play skills, symbolic play types and routines, and play level. This caregiver questionnaire measures play skill development over time. Increasing answers of "Yes" indicate growth in play skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No